CLINICAL TRIAL: NCT05026983
Title: Phase II Study of Binimetinib With Encorafenib in Patients With Metastatic Melanoma and CNS Metastases
Brief Title: Binimetinib and Encorafenib for the Treatment of Metastatic Melanoma and Central Nervous System Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0205; NCI-2021-08716 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0205 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-19; First posted 2021-08-30 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: conditions — Melanoma | interventions — binimetinib; encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (encorafenib, binimetinib) (Experimental): Patients receive encorafenib PO QD and binimetinib PO BID on day 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Encorafenib; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
Drug: Encorafenib — Given PO
  Other Names: Braftovi; LGX 818; LGX-818; LGX818
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effects of binimetinib and encorafenib in treating patients with melanoma that has spread to the central nervous system (metastases). Binimetinib and encorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving binimetinib and encorafenib may help control melanoma that has spread to the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate antitumor activity of high dosing regimen of encorafenib + binimetinib combination therapy for patients with BRAFV600-mutant melanoma brain metastases and/or leptomeningeal disease (LMD) as measured by progression free survival (PFS).

II. To evaluate the safety/tolerability of high dosing regimen of encorafenib + binimetinib combination therapy for patients with BRAFV600-mutant melanoma brain metastases and/or LMD.

SECONDARY OBJECTIVE:

I. To further evaluate antitumor activity of high dosing regimen of encorafenib + binimetinib combination therapy for patients with BRAFV600-mutant melanoma and/or LMD, as measured by brain metastasis response rate (BMRR), extracranial response rate, global response rate, brain metastases disease control rate (DCR), overall survival (OS), and duration of response (DOR).

EXPLORATORY OBJECTIVES:

I. To compare the immunological effects of this treatment on immune cells in the cerebrospinal fluid (CSF) to those observed in the peripheral blood.

II. To compare levels of encorafenib and binimetinib in the CSF and peripheral blood.

III. To assess neurocognitive function as measured by the Montreal Cognitive Assessment (MoCA) and MD Anderson Symptom Inventory brain tumor module (MDASI-BT).

OUTLINE:

Patients receive encorafenib orally (PO) once daily (QD) and binimetinib PO twice daily (BID) on day 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent.
* Age >= 18 years at the time of informed consent
* Histologically confirmed diagnosis of melanoma
* Presence of BRAFV600 mutation in tumor tissue previously determined by a local assay (including immunohistochemistry [IHC]) at any time prior to Screening or during Screening
* Cohort A: BRAF V600 mutant melanoma patients with progressive central nervous system (CNS) metastases. This includes patients with parenchymal brain metastases and/or LMD
* Cohort A: Prior therapy with Food and Drug Administration (FDA)-approved BRAF inhibitors (+/- MEK inhibitors) is required

  * No washout period is required
* Cohort A: Prior therapy with immunotherapy or other investigational agents is allowed

  * Washout period of 14 days since last dose
* Cohort B: BRAF V600 mutant melanoma patients who are treatment naive to BRAF/MEK inhibitors with CNS metastases, including LMD. Prior treatment with immunotherapy is permitted
* For patients with parenchymal brain metastases (mets) without LMD

  * Metastatic disease to the brain with at least 1 progressing parenchymal brain lesion >= 0.5 cm and =< 3 cm, defined as a magnetic resonance imaging (MRI) contrast-enhancing lesion that may be accurately measured in at least 1 dimension
* For patients with LMD

  * Patients must have investigator assessed radiographic and/or CSF cytological evidence of LMD
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of =< 2
* Patients may receive steroids to control symptoms related to CNS involvement

  * For patients with parenchymal brain metastases the dose must be =< 2 mg per 24 hours of dexamethasone (or the equivalent). Patient's symptoms should experience stability of neurological symptoms for at least 7 days, or on tapering dose of steroids. Physiologic replacement doses for adrenal insufficiency is allowed on this protocol
  * For patients with LMD: the dose must be =< 4 mg per 24 hours of dexamethasone (or the equivalent). Physiologic replacement doses for adrenal insufficiency is allowed on this protocol
* Radiation therapy:

  * For patients with parenchymal brain mets: prior radiation therapy, including stereotactic (SRS) or whole brain radiation (WBXRT) is allowed, but patient must be progressing in or having at least 1 new CNS lesion. Prior SBRT to extracranial lesions is allowed. Washout to prior radiation 14 days.
  * For patients with LMD: Patients who have received radiation to brain and/or spine, including WBXRT, SRS, or SBRT, are eligible, but must have completed radiation treatment at least 7 days prior to the start of treatment.
* Prior therapy with systemic immunotherapy or other investigational agents is allowed

  * Washout period of 14 days since last dose
* Other cancer directed treatment:

  * Concurrent treatment with other anti-cancer systemic therapies is not allowed. No other concomitant intrathecal therapy with another agent will be allowed. For patients that have received other systemic therapies, the minimum wash out period is as follows:

    * Patients that received previous intrathecal therapy must have received their last treatment >= 7 days prior to the start of treatment
    * Patients who have received systemic chemotherapy must have received their last treatment >= 21 days prior to the start of treatment

Patients must have appropriate laboratory parameters as defined below:

* Absolute neutrophil count (ANC) 1.5 X 10^9/L
* Hemoglobin 9.0 g/dL
* Platelets 75 X 10^9/L
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 X upper limit of normal (ULN)
* Total bilirubin =< 1.5 X ULN (isolated bilirubin > 1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)

  * NOTE: Patients with documented Gilbert syndrome or hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the primary investigator
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X ULN, in patients with liver metastases ≤5 X ULN
* Albumin ≥2.5 g/dL
* Creatinine ≤ 1.5 X ULN OR calculated creatinine clearance ≥50 mL/min OR 24-hour urine creatinine clearance ≥50 mL/min
* Female patients of childbearing potential must have a negative serum and/or urine pregnancy test result
* Female patients of childbearing potential must agree to protocol-approved methods of contraception and to not donate ova from Screening until 30 days after the last dose of study drug. Male patients must agree to use methods of contraception that are highly effective or acceptable and to not donate sperm from Screening until 90 days after the last dose of study drug
* The patient is deemed by the Investigator to have the initiative and means to comply with scheduled visits, treatment plan and study procedures

Exclusion Criteria:

* Evidence of active infection =< 7 days prior to initiation of study drug therapy (does not apply to viral infections that are presumed to be associated with the underlying tumor type required for study entry)
* Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 30 days of prior to study drug. Dead virus vaccines (e.g Flu) are allowed, even during treatment with study drug
* Inability to swallow and retain study treatment
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) even if fully immunocompetent on antiretroviral therapy (ART)
* Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to screening
  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2)
  * A left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition (MUGA) or echocardiogram (ECHO)
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia)
  * Baseline Fridericia's correction formula (QTcF) interval >= 480 msec. Can be repeated up to three times to confirm
* Concurrent neuromuscular disorder (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study treatment (e.g., uncontrolled nausea, vomiting or diarrhea; malabsorption syndrome; small bowel resection). Known history of acute or chronic pancreatitis
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease
* Use of herbal supplements, medications or foods that are moderate or strong inhibitors or inducers of cytochrome P450 (CYP) 3A4/5 =< 1 week prior to the start of study treatment
* History of a thromboembolic event < 12 weeks prior to starting study treatment. Examples of thromboembolic events include transient ischemia attack, cerebrovascular accident, deep vein thrombosis or pulmonary embolism. Catheter-related venous thrombosis is not considered a thromboembolic event for this trial even if < 12 weeks prior to starting study treatment. Note: Patients with either deep vein thrombosis or pulmonary emboli that do not result in hemodynamic instability are allowed to enroll as long as they are stable, asymptomatic and on stable anticoagulants for at least 2 weeks. Additionally, patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

  * NOTE: Patients with laboratory evidence of cleared HBV or HCV infection may be enrolled
  * NOTE: Patients with no prior history of HBV infection who have been vaccinated against HBV and who have a positive antibody against hepatitis B surface antigen as the only evidence of prior exposure may enroll
* Pregnancy or breastfeeding or patients who plan to become pregnant during the duration of the study
* Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Cohort A) | At 3 months
Incidence of dose-limiting toxicities (DLTs) | Up to 28 days
Incidence of adverse events (AEs) | Up to 30 days after last dose
  Graded according to the NCI CTCAE version 4.03 and changes in clinical laboratory parameters, vital signs, ECGs, ECHO/MUGA scans and ophthalmic examinations.
Incidence of dose interruptions, dose modifications and discontinuations due to AEs | Up to 3 years

SECONDARY OUTCOMES:
Progression free survival | From the date of first dose of study drug to the time of the first documented progression or death, whichever occurs first, assessed up to 3 years
Extracranial response rate | Up to 3 years
  Extracranial response rate is defined as the proportion of patients with a best overall extracranial response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 per investigator assessment.
Intracranial response rate | Up to 3 years
  Intracranial response rate is defined as the proportion of patients with a best overall Intracranial response of CR or PR according to modified (m)RECIST v1.1 per Investigator assessment. In addition, as part of our secondary endpoint, we will use Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria for response assessment.
Disease control rate | Up to 3 years
  Defined as the proportion of patients with a best overall response of CR, PR or stable disease (SD) per Investigator assessment.
Duration of response (DOR) | From first documented response of CR or PR per Investigator assessment until first documented progression or death due to any cause, whichever occurs first, assessed up to 3 years
  DOR will be estimated using the Kaplan-Meier method. DOR estimates along with two-sided 95% confidence interval is will be presented.
Overall survival (OS) | From the date of first dose of study drug to the date of death due to any cause, assessed up to 3 years
  The survival distribution function for OS will be estimated using the Kaplan-Meier method. OS estimates along with two-sided 95% Cis will be presented. Associations between OS and demographic/clinical measures may be evaluated using Cox proportional hazards regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Isabella C Glitza, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Corradi G, De Martino S, Rinaldi A, Siepe G, Marchese PV, Melotti B, Comito F. Rapid radiological response of leptomeningeal carcinosis and prolonged survival to encorafenib and binimetinib in BRAF-mutated melanoma. Anticancer Drugs. 2025 Sep 1;36(8):691-693. doi: 10.1097/CAD.0000000000001737. Epub 2025 May 30. PMID 40439484
- See also: M D Anderson Cancer Center — http://www.mdanderson.org